CLINICAL TRIAL: NCT05909683
Title: A Randomized Prospective Clinical Trial to Assess Procalcitonin-guidance and Molecular-guided Diagnosis as Mainstay for Therapy of Severe Infections (the MODIFY Trial)
Brief Title: Assessing the Procalcitonin-guidance and Molecular-guided Diagnosis for Therapy of Severe Infections (the MODIFY Trial)
Acronym: MODIFY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MODIFY; 2022-502962-26-00 (Other: EMA CTIS)
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Sepsis
Keywords: Severe infections; Antibiotics; Procalcitonin; Blood Culture Identification 2 Panel (BCID2); Reveal Rapid AST system
MeSH Terms: conditions — Sepsis; Infections | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: According to protocol study intervention is not study drug administration; intervention includes two steps: modification of antibiotics administered; duration of antibiotic treatment. SOC patients will receive antibiotics according to standard practice of the attending physicians.
  MODIFY strategy group patients will start antibiotics according to standard practice. They will be informed after randomization about the results of BCID2, Reveal Rapid AST and PCT. Physicians and investigators receiving this information are obliged to change the empirically prescribed antibiotics (escalate, de- escalate or stop) aiming to improve patient outcomes. Exceptions to overrule this algorithm will be accepted for medically unstable patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-care (Sham Comparator): These patients will receive antibiotics according to standard practice of the attending physicians. The central lab will feedback to attending physicians and investigators the results of the conventional blood cultures and AST according to the routine SOP. The attending physicians and investigators will be allowed to decide for any change of antimicrobial treatment based on the results of conventional blood cultures provided to them by the central lab or any other culture provided to them by their hospital. Antibiotics will be stopped according to the local standard practice. BCID2, Reveal Rapid AST and PCT will be performed in the samples of these patients, attending physicians will not be provided such information.
  Interventions: Other: Standard of Care
- MODIFY strategy (Experimental): These patients will start antibiotics according to standard practice of the attending physicians. It is anticipated that attending physicians will be informed in maximum 5 hours after randomization about the results of BCID2 including carriage of resistance genes and of the Reveal Rapid AST in the case of Gram-negative isolates. Physicians and investigators receiving this information are obliged to change the empirically prescribed antibiotics according to the rule provided in Box 1. The attending physicians and investigators will be allowed to decide for any change of antimicrobial treatment based on the results of conventional blood cultures provided to them by the central lab or any other culture provided to them by their hospital. PCT will be measured on day 1 and then daily starting from day 5. Attending physicians will be advised to discontinue antimicrobials on the first day by day 5 when PCT value is less than 80% of the initial value or it remains below 0.5 ng/ml.
  Interventions: Diagnostic Test: Change of antimicrobials based on BCID2 and Reveal Rapid AST tests. Stop of antimicrobials based on PCT results.

INTERVENTIONS:
Diagnostic Test: Change of antimicrobials based on BCID2 and Reveal Rapid AST tests. Stop of antimicrobials based on PCT results. — After the patient's blood flask is flagged positive for bloodstream infection, the blood sample will be assessed in the BCID2 diagnostic test in order to identify the underlying pathogens the patient is infected with. After the identification, and in the presence of gram-negative bacteria, the sample will be assessed in the Reveal Rapid AST test to provide information about which antimicrobials the specific pathogens are sensitive to. When both the identification of the pathogen and the sensitivities are available, the central laboratory will inform the attending physicians, who are obliged to change the standard of care antimicrobial therapy administered based on the rule in Box1 of the protocol. Finally, based on the results of the procalcitonin (PCT) on the first day by day 5 when PCT value is less than 80% of the initial value or it remains below 0.5 ng/ml, the attending physicians should discontinue the antimicrobial therapy.
  Arms: MODIFY strategy
Other: Standard of Care — Standard of care practices of the specific study site. Antimicrobials will be administered based on the attending physicians' critical opinion, and discontinuation will be done based on the standard procedures of the study site.
  Arms: Standard-of-care

SUMMARY:
MODIFY is a randomized, open-labeled, and prospective study that will be conducted in multiple Intensive Care Units (ICUs) and departments of Internal Medicine across Greece. It aims to change the traditional approach for the management of severe infections by integrating the results of BCID2, Reveal Rapid AST, and PCT, to improve patients' outcomes. Early and precise identification of the underlying causative pathogen along with the fast acquisition of the antimicrobial sensitivity results may positively impact the uncontrolled antimicrobial prescription.

DETAILED DESCRIPTION:
Early administration of antimicrobials remains the mainstay of treatment of severe infections. The time until start of antimicrobials is so crucial that every hour of delay impacts considerably on mortality. In everyday clinical practice even when antimicrobials are administered early, it is impossible to know whether they are appropriate or not because cultures of specimens collected from the patient require at least 48 to 72 hours to provide some information about the type of pathogen and the antimicrobial susceptibilities.

BioFire ® FilmArray ® possesses four Food and Drug Administration (FDA)-cleared panels of molecular diagnosis, capable of detecting multiple targets in less than an hour of sample handling. Among them, Blood Culture Identification 2 Panel (BCID2) covers 43 targets. BCID2 provides information on the genes of resistance to antibiotics the microorganisms carry. BCID2 combined with fast AST can, however, introduce revolutionary changes in minimizing the time until the appropriate antimicrobial is prescribed. The concept of Reveal is to provide AST for a full panel of antibiotics if one Gram-negative isolate is identified in the blood flask.

Evaluation of the appropriateness of the administered therapy and decision about discontinuation or de-escalation of antimicrobials, is based on the use of biomarkers and mainly procalcitonin (PCT).

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* For women of child-bearing potential, willingness to avoid pregnancy during the study and agreement to notify investigator if pregnancy occurs.
* Age more than or equal to 18 years
* Patients who have completed their participation in another study for more than 30 days can be included in this study.
* Written informed consent provided by the patient or by their legal representative in case of patients unable to consent due to sepsis onset affecting their mental capacity.
* Sepsis defined by the Sepsis-3 definition; this is defined separately for community-acquired sepsis and for hospital-acquired sepsis. Community-acquired sepsis is defined as any SOFA score 2 points or more for patients admitted in hospital emergencies with community-acquired pneumonia (CAP), community-acquired acute pyelonephritis (AP) or community-acquired primary bacteremia (BSI). CAP, AP and BSI are considered community-acquired for patients who have no history of hospitalization lasting more than 2 days the last 90 days or who are not under hemodialysis or who are not residents of long-term care facilities. Hospital-acquired sepsis is defined as any SOFA score increase by 2 points or more from the admission SOFA score for patients with onset of hospital-acquired pneumonia (HAP), ventilator-associated pneumonia (VAP), acute pyelonephritis (AP) or primary bacteremia (BSI) at least 48 hours after hospital admission. For patients with history of hospitalization lasting more than 2 days the last 90 days or who are under hemodialysis or who are residents of long-term care facilities and are admitted to hospital with HAP, VAP, AP and BSI the definition of hospital-acquired sepsis applies. In this case, the baseline SOFA score is considered as the known SOFA score before infection onset.
* Presence of one of the following infections: community-acquired pneumonia (CAP), hospital-acquired pneumonia (HAP), ventilator-associated pneumonia (VAP), acute pyelonephritis (AP) and primary bacteremia (BSI).
* Positive blood culture

Exclusion Criteria:

* Failure to obtain written consent to participate
* Previous enrollment in this study within the past 90 days. Patients enrolled in another study will not be accepted.
* Patients in pregnancy or breastfeeding. Women of child-bearing potential will be screened by a urine pregnancy test before inclusion in the study
* Patients receiving prolonged antibiotic therapies (e.g. endocarditis, implantable device-associated infection, cerebral/hepatic abscess, osteomyelitis, meningitis)
* Patients with severe infections due to viruses or parasites (e.g. Dengue, Toxoplasma gondii, Plasmodium spp.)
* Patients with infection due to Mycobacterium tuberculosis.
* Patients suffering from cystic fibrosis
* Severely immunocompromised patients such as a) patients with infection by the human immunodeficiency virus and with a CD4 count of less than 200 cells/mm3; b) neutropenic patients with less than 500 neutrophils/mm3; and c) patients with solid organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
The number of days under treatment with broad-spectrum antibiotics in the group receiving the MODIFY strategy compared to patients treated by standard of care. | Through study completion, an average of 2 years
  The number of days under treatment with broad-spectrum antibiotics in the group receiving the MODIFY strategy compared to patients treated by standard of care.

SECONDARY OUTCOMES:
Time to first change of antimicrobial modification | Through study completion, an average of 2 years
  Time to first change of antimicrobial modification
Time to the first sterile blood culture | Through study completion, an average of 2 years
  Time to the first sterile blood culture
The number of patients in whom no changes in administered antibiotics will apply. | Through study completion, an average of 2 years
  The number of patients in whom no changes in administered antibiotics will apply.
At least 2-point decrease of baseline SOFA (Sequential organ failure assessment) score by day 7 | Through study completion, an average of 2 years
  At least 2-point decrease of baseline SOFA (Sequential organ failure assessment) score by day 7. SOFA ranges between 0-24 and the higher the score, the worst the outocome of the patient.
28-day mortality | Through study completion, an average of 2 years
  28-day mortality
90-day mortality | Through study completion, an average of 2 years
  90-day mortality
Incidence of laboratory documented Clostrioides difficile infection | Through study completion, an average of 2 years
  Incidence of laboratory documented Clostrioides difficile infection
Length of hospital stay | Through study completion, an average of 2 years
  Length of hospital stay
Cost of hospitalization | Through study completion, an average of 2 years
  Cost of hospitalization
Time to escalation of antibiotics | Through study completion, an average of 2 years
  Time to escalation of antibiotics
Time to de-escalation of antibiotics | Through study completion, an average of 2 years
  Time to de-escalation of antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giamarellos-Bourboulis, MD,PhD, Study Chair — Hellenic Institute for the Study of Sepsis
Locations (15):
- Greece (15):
  - Intensive Care Unit of Center for Respiratory Failure, Sotiria Chest Diseases Athens General Hospital, Athens, Attica
  - New Multivalent Intensive Care Unit, Sotiria Chest Diseases Athens General Hospital, Athens, Attica
  - 2nd Propaedeutic Department of Internal Medicine, Attikon University Hospital, Athens, Chaidari
  - 4th Department of Internal Medicine, Attikon University Hospital, Athens, Chaidari
  - 1st Department of Internal Medicine, General Hospital of Elefsina "Thriasio", Athens, Elefsina
  - 2nd Department of Internal Medicine, University General Hospital of Alexandroupolis, Alexandroupoli
  - 1st Department of Internal Medicine, General Hospital of Athens KORGIALENIO-BENAKIO E.E.S., Athens
  - 1st Department of Internal Medicine- General Hospital of Athens GENNIMATAS, Athens
  - 3rd University Department of Internal Medicine, Sotiria Athens General Hospital, Athens
  - 1st Department of Internal Medicine - General Hospital of Athens Sismanoglio- Amalia Fleming, Athens
  - 3rd Department of Internal Medicine - General State Hospital of Nikaia "Saint Panteleimon" - West Attica General Hospital "Agia Varvara", Athens
  - Clinic of Intensive Care and Pulmonary Diseases, Aghioi Anargyroi Kifissia General Oncologic Hospital, Kifissia
  - 2nd Department of Internal Medicine, General Hospital of Piraeus "Tzaneio", Piraeus
  - 1st University Department of Internal Medicine, AHEPA University General Hospital of Thessaloniki, Thessaloniki
  - Intensive Care Unit, Ippokrateion General Hospital, Thessaloniki